CLINICAL TRIAL: NCT01862276
Title: Role of Bile Duct Resection in Major Hepatectomy Due to Intrahepatic Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: KHBO1206; UMIN000010416 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-05-14; First posted 2013-05-24 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate the prognosis due to presence or absence of bile duct resection in intrahepatic cholangiocarcinoma that require hepatic lobectomy.

DETAILED DESCRIPTION:
The bile duct resection in hepatic lobectomy due to cholangiocarcinoma, mass forming type, is still controversial. We retrospectively evaluated the effect of bile duct resection in this surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cases of major hepatectomy due to intrahepatic cholangiocarcinoma

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent hepatic lobectomy between 2000 and 2010 for intrahepatic cholangiocarcinoma, and did not undergo adjuvant chemotherapy will be included for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
3-year recurrence-free survival rate | 11 years (2000-2010)
Ratio of local recurrence at the hepatico-duodenal ligament | 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Nagano, MD, PhD, Study Director — Osaka University Graduate School of Medicine
Locations (1):
- Osaka University, Graduate School of Medicine, Osaka, Osaka, Japan